CLINICAL TRIAL: NCT02453672
Title: A Randomised, Double-blind, Three-arm, Parallel Group, Single-dose Study to Compare the Pharmacokinetics, Safety, Tolerability, and Immunogenicity of Three Formulations of Bevacizumab (SB8, EU Sourced Avastin®, and US Sourced Avastin®) in Healthy Male Subjects
Brief Title: Pharmacokinetic, Safety, Tolerability, and Immunogenicity Study of SB8 in Healthy Male Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Samsung Bioepis Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: SB8-G11-NHV; 2015-001026-41 (EudraCT Number)
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Results first posted 2019-06-03 (Actual); Last update posted 2019-06-03 (Actual); Status verified 2019-02

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- SB8 (Experimental): SB8, single dose of 3 mg/kg, IV infusion
  Interventions: Biological: SB8
- EU Sourced Avastin® (Active Comparator): EU Sourced Avastin®, single dose of 3 mg/kg, IV infusion
  Interventions: Biological: EU sourced Avastin®
- US Sourced Avastin® (Active Comparator): US Sourced Avastin®, single dose of 3 mg/kg, IV infusion
  Interventions: Biological: US Sourced Avastin®

INTERVENTIONS:
Biological: SB8 — SB8, proposed bevacizumab biosimilar
  Arms: SB8
Biological: EU sourced Avastin® — EU sourced Avastin® (bevacizumab, Roche Registration Ltd.)
  Arms: EU Sourced Avastin®
Biological: US Sourced Avastin® — US Sourced Avastin® (bevacizumab, Roche Registration Ltd.)
  Arms: US Sourced Avastin®

SUMMARY:
Pharmacokinetics, Safety, Tolerability, and Immunogenicity of Three Formulations of Bevacizumab

DETAILED DESCRIPTION:
A Randomised, Double-blind, Three-arm, Parallel Group, Single-dose Study to Compare the Pharmacokinetics, Safety, Tolerability, and Immunogenicity of Three Formulations of Bevacizumab (SB8, EU Sourced Avastin®, and US Sourced Avastin®) in Healthy Male Subjects

ELIGIBILITY:
Inclusion Criteria:

* Healthy male subjects
* Have body weight between 65.0-90.0 kg (inclusive) and body mass index between 20.0-29.9 kg/m2 (inclusive)

Exclusion Criteria:

* Have a history of hypersensitivity or allergic reactions to bevacizumab or to any of the excipients
* Have a history of and/or current clinically significant gastrointestinal, renal, hepatic, cardiovascular, haematological, pulmonary, neurologic, metabolic, psychiatric, or allergic disease excluding mild asymptomatic seasonal allergies
* Have a history of arterial thromboembolic events including cerebrovascular accidents, transient ischaemic attacks, and myocardial infarction
* Have a history of and/or current cardiac disease
* Have previously been exposed to vascular endothelial growth factor (VEGF) antibody, any other antibody, or protein targeting the VEGF receptor
* Have a history of cancer including lymphoma, leukaemia, and skin cancer.
* Have received live vaccine(s) within 30 days prior to Screening visit or who will require a vaccine(s) between Screening and the end of study visit
* Have taken medication with a half-life of > 24 hours within 30 days or 10 half-lives of the medication prior to the IP administration

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 119 (Actual)
Dates: Start 2015-04; Primary Completion 2015-09 (Actual); Study Completion 2015-09 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Samsung Investigational Site, Antwerp, Belgium

REFERENCES:
- [Derived] Shin D, Lee YJ, Choi J, Lee D, Park M, Petkova M. A phase I, randomized, single-dose pharmacokinetic study comparing sb8 (bevacizumab biosimilar) with reference bevacizumab in healthy volunteers. Cancer Chemother Pharmacol. 2020 Oct;86(4):567-575. doi: 10.1007/s00280-020-04144-7. Epub 2020 Sep 19. PMID 32949267

RESULTS

PARTICIPANT FLOW:
Groups:
- SB8 (Proposed Bevacizumab Biosimilar): SB8, single dose of 3 mg/kg, IV infusion
  SB8: SB8, proposed bevacizumab biosimilar
Period: Overall Study
Arm/Group | SB8 (Proposed Bevacizumab Biosimilar) | EU Sourced Avastin® | US Sourced Avastin®
Started | 40 | 40 | 39
Completed | 37 | 38 | 38
Not Completed | 3 | 2 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | SB8 (Proposed Bevacizumab Biosimilar) | EU Sourced Avastin® | US Sourced Avastin® | Total
Number analyzed (Participants) | 40 | 40 | 39 | 119
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.2 (9.24) | 39.5 (10.45) | 38.9 (9.32) | 40.9 (9.90)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0 | 0
  Male | 40 | 40 | 39 | 119

OUTCOME MEASURES:

1. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to Infinity (AUCinf)
Description: 0 (pre-dose), 0.75, 1.5 (end of infusion), 3, 6, 12, 24, 48, and 96 hours, then at Day 8 (168 h), 15 (336 h), 22 (504 h), 29 (672 h), 43 (1008 h), 57 (1344 h), 71 (1680 h), and 85 (2016 h) after start of infusion.
Time Frame: 0 to 2016 hours after start of infusion
Population: Among the subjects discountinued, subjects with major protocol deviations were excluded from the PK population for the PK analysis.
Measure: Mean (Standard Deviation); unit: h·μg/mL
Arm/Group | SB8 (Proposed Bevacizumab Biosimilar) | EU Sourced Avastin® | US Sourced Avastin®
Number analyzed (Participants) | 38 | 38 | 38
h·μg/mL | 25354.4 (4833.10) | 28896.8 (6221.62) | 28684.8 (5425.14)

2. Primary Outcome: Area Under the Concentration-time Curve From Time Zero to the Last Quantifiable Concentration (AUClast)
Description: as for outcome 1
Time Frame: 0 to 2016 hours after start of infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h·μg/mL
Arm/Group | SB8 (Proposed Bevacizumab Biosimilar) | EU Sourced Avastin® | US Sourced Avastin®
Number analyzed (Participants) | 38 | 38 | 38
h·μg/mL | 24199.2 (4367.53) | 27342.2 (5374.53) | 27177.9 (4770.93)

3. Primary Outcome: Maximum Serum Concentration (Cmax)
Description: as for outcome 1
Time Frame: 0 to 2016 hours after start of infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: μg/mL
Arm/Group | SB8 (Proposed Bevacizumab Biosimilar) | EU Sourced Avastin® | US Sourced Avastin®
Number analyzed (Participants) | 38 | 38 | 38
μg/mL | 76.259 (14.6999) | 76.059 (11.7053) | 76.485 (16.9916)

4. Secondary Outcome: Time to Reach Cmax (Tmax)
Description: as for outcome 1
Time Frame: 0 to 2016 hours after start of infusion
Population: as for outcome 1
Measure: Mean (Standard Deviation); unit: h
Arm/Group | SB8 (Proposed Bevacizumab Biosimilar) | EU Sourced Avastin® | US Sourced Avastin®
Number analyzed (Participants) | 38 | 38 | 38
h | 3.639 (2.1885) | 3.638 (2.4261) | 5.646 (15.6665)

ADVERSE EVENTS:
Time Frame: 12 weeks
Arm/Group | SB8 (Proposed Bevacizumab Biosimilar) | EU Sourced Avastin® | US Sourced Avastin®
All-Cause Mortality (participants affected / at risk) | 0/40 | 0/40 | 0/39
Serious Adverse Events (participants affected / at risk) | 1/40 | 0/40 | 0/39
Other Adverse Events (participants affected / at risk) | 20/40 | 15/40 | 21/39
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SB8 (Proposed Bevacizumab Biosimilar) (N=40) | EU Sourced Avastin® (N=40) | US Sourced Avastin® (N=39)
Perirectal abscess (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | SB8 (Proposed Bevacizumab Biosimilar) (N=40) | EU Sourced Avastin® (N=40) | US Sourced Avastin® (N=39)
Diarrhoea (Gastrointestinal disorders) | 4 | 2 | 0
Abdominal discomfort (Gastrointestinal disorders) | 2 | 0 | 0
Haemorrhoids (Gastrointestinal disorders) | 1 | 0 | 0
Nausea (Gastrointestinal disorders) | 1 | 0 | 0
Toothache (Gastrointestinal disorders) | 1 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0
Abdominal pain (Gastrointestinal disorders) | 0 | 1 | 1
Stomatitis (Gastrointestinal disorders) | 0 | 0 | 1
Influenza like illness (General disorders) | 1 | 0 | 0
Fatigue (General disorders) | 0 | 2 | 0
Catheter site pain (General disorders) | 0 | 0 | 1
Chest pain (General disorders) | 0 | 0 | 1
Nasopharyngitis (Infections and infestations) | 3 | 6 | 6
Conjunctivitis (Infections and infestations) | 0 | 0 | 1
Oral herpes (Infections and infestations) | 0 | 0 | 1
Otitis externa (Infections and infestations) | 0 | 1 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0
Ligament sprain (Injury, poisoning and procedural complications) | 0 | 0 | 1
Rib fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Back pain (Musculoskeletal and connective tissue disorders) | 2 | 1 | 2
Myalgia (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Neck pain (Musculoskeletal and connective tissue disorders) | 1 | 0 | 1
Muscle spasms (Musculoskeletal and connective tissue disorders) | 1 | 0 | 0
Musculoskeletal stiffness (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1
Headache (Nervous system disorders) | 3 | 0 | 7
Somnolence (Nervous system disorders) | 1 | 0 | 1
Syncope (Nervous system disorders) | 0 | 0 | 1
Dysuria (Renal and urinary disorders) | 0 | 1 | 1
Erectile dysfunction (Reproductive system and breast disorders) | 1 | 0 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 2 | 0 | 2
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 1
Erythema (Skin and subcutaneous tissue disorders) | 1 | 0 | 1
Acne (Skin and subcutaneous tissue disorders) | 0 | 1 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes